CLINICAL TRIAL: NCT01735227
Title: Single-center Randomized Controlled Study of Omeprazole and Pantoprazole Antiplatelet Effect of Clopidogrel Clinical Randomized Controlled Trials
Brief Title: Omeprazole and Pantoprazole Antiplatelet Effect of Clopidogrel Clinical Trials(OPEN)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yaling Han (Other)
Responsible Party: Sponsor-Investigator, Yaling Han, vice president, Shenyang Northern Hospital
Organization: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NH2012-9-20
Record Dates: First submitted 2012-11-14; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Acute Coronary Syndromes
Keywords: pantoprazole; omeprazole; anti - platelet effect
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Omeprazole; Pantoprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omeprazole group (Experimental): omeprazole group:all patients taking clopidogrel loading dose 300mg + aspirin 300mg and the subsequent maintenance dose of clopidogrel 75mg(1 year) + aspirin 300mg(1 month)+ aspirin 100mg(long-term)and taking omeprazole 20mg/d(1 month).on the day of admission ( before medication ) , medication for 12-24 hours , medication after 72 hours , 30 days , each taken early morning fasting venous blood again , measuring AA 、ADP - induced platelet aggregation . And selected 30 days , 6 months and 12 months to record the patient's clinical adverse events ( including death , myocardial infarction , and any revascularization , stent thrombosis , recurrent angina , rehospitalization due to cardiovascular disease , bleeding events) .
  Interventions: Drug: omeprazole; Drug: Pantoprazole
- pantoprazole group (Experimental): pantoprazole group: all patients taking clopidogrel loading dose 300mg + aspirin 300mg and the subsequent maintenance dose of clopidogrel 75mg(1 year) + aspirin 300mg(1 month)+ aspirin 100mg(long-term),taking pantoprazole 20mg/d(1 month).
  Interventions: Drug: omeprazole; Drug: Pantoprazole

INTERVENTIONS:
Drug: omeprazole — all patients taking clopidogrel loading dose 300mg + aspirin 300mg and the subsequent maintenance dose of clopidogrel 75mg(1 year) + aspirin 300mg(1 month)+ aspirin 100mg(long-term)and omeprazole group taking omeprazole 20mg/d
Drug: Pantoprazole — On the day of admission , all patients taking clopidogrel loading dose 300mg + aspirin 300mg and the subsequent maintenance dose of clopidogrel 75mg + aspirin 300mg and omeprazole group taking omeprazole 20mg / d , pantoprazole group taking pantoprazole 20mg / d. Respectively, on the day of admission ( before medication ) , medication for 12-24 hours , medication after 72 hours , 30 days , each taken early morning fasting venous blood again , measuring AA 、ADP - induced platelet aggregation . And selected 30 days , 6 months and 12 months to record the patient's clinical adverse events ( including death , myocardial infarction , and any revascularization , stent thrombosis , recurrent angina , rehospitalization

SUMMARY:
In order to further clarify the interaction of PPIs with clopidogrel anti - platelet effect , the investigators designed a clinical randomized controlled trials of omeprazole and pantoprazole antiplatelet effect of clopidogrel .In this experiment , the investigators have taken a randomized NSTE-ACS hospitalized patients met the inclusion criteria were randomly divided into omeprazole and pantoprazole groups . On the day of admission , all patients taking clopidogrel loading dose 300mg + aspirin 300mg and the subsequent maintenance dose of clopidogrel 75mg + aspirin 300mg and omeprazole group taking omeprazole 20mg / d , pantoprazole group taking pantoprazole 20mg / d. Respectively, on the day of admission ( before medication ) , medication for 12-24 hours , medication after 72 hours , 30 days , each taken early morning fasting venous blood again , measuring AA 、ADP - induced platelet aggregation . And selected 30 days , 6 months and 12 months to record the patient's clinical adverse events ( including death , myocardial infarction , and any revascularization , stent thrombosis , recurrent angina , rehospitalization due to cardiovascular disease , bleeding events) . To assess the impact of PPIs on clopidogrel antiplatelet effect by observing 1 year follow-up results , and further explore the optimal combination of dual anti-platelet and joint PPIs course of treatment , appropriate dosage and the best time to provide reasonable for clinical programs to create a personalized treatment system , improve the patient's quality of life .

DETAILED DESCRIPTION:
Through a number of large-scale clinical trials , Meta analysis, and clinical treatment guidelines confirm that clopidogrel and aspirin dual antiplatelet treatment strategies for acute coronary syndrome (ACS) undergoing percutaneous coronary interventions(PCI) of stent implantation surgery patients have a vital role . It can effectively suppress acute 、subacute stent thrombosis formation , reduce readmissions ratio , thus greatly improving the quality of life of patients . A large number of clinical practice reports, although the treatment strategies to reduce the incidence of adverse cardiovascular events ,it has increased the possibility of the occurrence of gastrointestinal bleeding complications . Proton pump inhibitors (PPIs) are often used to prevent gastrointestinal complications of dual antiplatelet therapy . 2008 American College of Cardiology (ACC) / American Society of Gastroenterology (ACG) / American Heart Association (AHA) jointly issued a consensus document , consistently recommended that the majority of clinicians application of dual antiplatelet and PPIs treatment for patients with risk factors for gastrointestinal bleeding that may exist at the same time ,in order to reduce the occurrence of gastrointestinal adverse events . But at home and abroad in recent years, there have been reports suggest that the interaction of PPIs with clopidogrel may exist , thereby reduce the latter 's anti- platelet effect , in order to make the incidence of adverse CV events increased about 25-64 % . In January 2009 , the U.S. Food and Drug Administration (FDA) announced a safety review of an earlier report on the potential interaction of these two types drugs , particularly stressed the need to carry out a large number of clinical practice research further to clear both the interaction . PPIs antiplatelet effects of clopidogrel after PCI is not yet very clear , clinical results on both interactions still exist many different academic perspectives and research defects , so still need to arouse sufficient attention , continue to carry out the relevant fields research .

In order to further clarify the interaction of PPIs with clopidogrel anti - platelet effect , the investigators designed a clinical randomized controlled trials of omeprazole and pantoprazole antiplatelet effect of clopidogrel .In this experiment , the investigator have taken a randomized NSTE-ACS hospitalized patients met the inclusion criteria were randomly divided into omeprazole and pantoprazole groups . On the day of admission , all patients taking clopidogrel loading dose 300mg + aspirin 300mg and the subsequent maintenance dose of clopidogrel 75mg + aspirin 300mg and omeprazole group taking omeprazole 20mg / d , pantoprazole group taking pantoprazole 20mg / d. Respectively, on the day of admission ( before medication ) , medication for 12-24 hours , medication after 72 hours , 30 days , each taken early morning fasting venous blood again , measuring AA 、ADP - induced platelet aggregation . And selected 30 days , 6 months and 12 months to record the patient's clinical adverse events ( including death , myocardial infarction , and any revascularization , stent thrombosis , recurrent angina , rehospitalization due to cardiovascular disease , bleeding events) . To assess the impact of PPIs on clopidogrel antiplatelet effect by observing 1 year follow-up results , and further explore the optimal combination of dual anti-platelet and joint PPIs course of treatment , appropriate dosage and the best time to provide reasonable for clinical programs to create a personalized treatment system , improve the patient's quality of life .

ELIGIBILITY:
Inclusion Criteria:

1. ACS (including unstable angina pectoris, non-ST-segment elevation myocardial infarction and ST-elevation myocardial infarction) ;
2. The age between18 and 75 ;
3. Informed consent.

Exclusion Criteria:

1. Receiving GP IIb / IIIa receptor antagonist treatment;
2. Had received prior to enrollment 7d cilostazol;
3. Dual antiplatelet therapy contraindications;
4. NYHA grade III ~ IV;
5. Presence of multivessel severe coronary lesions , need elective coronary revascularization;
6. The need for long-term use of warfarin after valve surgery or persistent atrial fibrillation;
7. Severe liver or kidney dysfunction;
8. Has not been cured of peptic ulcer or presence of bleeding tendency;
9. Who complicate the known bleeding tendency and blood system diseases;
10. Have a history of intracranial hemorrhage within 6 monhs;
11. Planned surgery recently;
12. Pregnancy;
13. Other serious illness, life expectancy less than 6 months;
14. Nearly 1 year underwent PCI , regular take aspirin 、clopidogrel since;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Platelet aggregation rate(AA 、ADP) | 30 days

SECONDARY OUTCOMES:
clinical adverse events | 12 months
  1. MACE(including cardiac death, acute myocardial infarction , target lesion revascularization , shock);
  2. stent thrombosis;
  3. stroke

CONTACTS AND LOCATIONS:
Overall Officials: Han Yaling, MD, Principal Investigator — Shenyang Northern Hospital
Locations (2):
- China (2):
  - OPEN trail, Shenyang, Liaoning
  - ShenyangNH, Shenyang, Liaoning

REFERENCES:
- [Derived] Gu RX, Wang XZ, Li J, Deng J, Li XX, Wang J. Effects of omeprazole or pantoprazole on platelet function in non-ST-segment elevation acute coronary syndrome patients receiving clopidogrel. Mil Med Res. 2016 Dec 15;3:38. doi: 10.1186/s40779-016-0107-0. eCollection 2016. PMID 28018669